CLINICAL TRIAL: NCT06455839
Title: Breathwork Intervention for Individuals With Chronic Musculoskeletal Pain
Brief Title: Breathwork for Chronic Musculoskeletal Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Adam Hanley, Principal Investigator, Florida State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00005048
Record Dates: First submitted 2024-06-07; First posted 2024-06-12 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Pain; Chronic Pain; Pain, Chronic; Musculoskeletal Pain
MeSH Terms: conditions — Pain; Chronic Pain; Musculoskeletal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Guided Respiration Mindfulness Therapy (Experimental)
  Interventions: Behavioral: Guided Resipiration Mindfulness Therapy (GRMT)

INTERVENTIONS:
Behavioral: Guided Resipiration Mindfulness Therapy (GRMT) — GRMT provides training in respiratory regulation, mindfulness and relaxation. The GRMT training will begin with a 15-minute introduction to the treatment model, followed by an hour of therapist-guided respiration (i.e., continuous rhythmic expansion of the chest, and relaxed exhalation involving release of all respiratory and peripheral musculature). The final 45 minutes will be used to discuss participant experiences during the GRMT training. GRMT training sessions will occur in-person and in a small group format (<5 participants each).

SUMMARY:
This project is a single-site, single-arm, clinical feasibility trial examining the impact of a single-session, 2-hour connected consciousness breathing with breath retention (CCBR) training for chronic musculoskeletal pain.

DETAILED DESCRIPTION:
CCBR is a breathwork style that involves breathing with no pause between inhalation and exhalation (also known as circular breathing). This breathing pattern is maintained for a given period of time, ranging from 5 minutes to over 2 hours. In the proposed project, the CCBR training will begin with a 15-minute introduction to CCBR, followed by an hour and 15 minutes of therapist-guided CCBR practice. The final 30 minutes will be used to discuss participant experiences during the CCBR practice. CCBR training sessions will occur in-person and in a small group format (5 participants each).

ELIGIBILITY:
Inclusion Criteria:

* having received a professional diagnosis of clinical levels of chronic pain
* being able to not commit to another (new) treatment during the course of the study
* understanding English instructions fluently
* Being 18 and above

Exclusion Criteria:

* having learned to practice breathwork any time in the past
* being unable to perform most basic tasks due to pain or pain treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-05-29 (Actual); Primary Completion 2024-06-11 (Actual); Study Completion 2024-07-27 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Chronic Pain Recruited | 1 week
  Examine recruitment rates during the 1 week of recruitment.
Intervention Adherence | 2 Hours
  Examine the percentage of participants completing their 2-hour intervention session.
Treatment Acceptability | Completed immediately after the 2-hour GRMT training
  Treatment acceptability will be assessed with a 12-item adaptation of the Treatment Framework of Acceptability questionnaire. Scores range from 5 to 45. Higher scores reflect greater acceptability.

SECONDARY OUTCOMES:
Global Impression of Change | Completed at 2- and 6-week follow-ups
  Treatment related improvement will be assessed with the Patient Global Impression of Change scale. Scores range from 0 to 7, with higher scores reflecting greater treatment related improvement.

OTHER OUTCOMES:
Acute Pain Unpleasantness | Will be completed immediately before and after the 2-hour intervention session
  Change in acute pain unpleasantness will be measured with an individual item ("How unpleasant is your pain, right now?") rated on a numeric rating scale. Scores range from 0 to 10, with higher scores reflecting greater acute pain unpleasantness.
Acute Pain Intensity | Will be completed immediately before and after the 2-hour intervention session
  Change in acute pain intensity will be measured with an individual item ("How much pain do you have, right now?") rated on a numeric rating scale. Scores range from 0 to 10, with higher scores reflecting greater acute pain intensity.
Daily Pain Intensity | Daily for 6 weeks
  Change in daily pain intensity from from the first post-intervention day through the 6-week follow-up will be assessed with the pain intensity item from the Pain, Enjoyment, and General Activity scale. Scores range from 0 to 10, with higher scores reflecting greater pain intensity.
Daily Pain Interference | Daily for 6 weeks
  Change in daily pain interference from from the first post-intervention day through the 6-week follow-up will be assessed with the two pain interference items from the Pain, Enjoyment, and General Activity scale. Scores range from 0 to 10, with higher scores reflecting greater pain interference.
Chronic Pain | Baseline, 2 weeks post-treatment, 6 week post-treatment
  Change in chronic pain from baseline through 6-week follow-up will be assessed with the Pain, Enjoyment, and General Activity scale. Scores range from 0 to 10, with higher scores reflecting greater chronic pain.
Sleep | Baseline, 2 weeks post-treatment, 6 week post-treatment
  Change in sleep from baseline through 6-week follow-up will be assessed with the PROMIS Sleep Disturbance Short Form. Scores range from 6 to 30, with higher scores reflecting worse sleep.
Pain Catastrophizing | Baseline, 2 weeks post-treatment, 6 week post-treatment
  Change in pain catastrophizing from baseline through 6-week follow-up will be assessed with the Pain Catastrophizing Scale. Scores range from 0 to 52, with higher scores reflecting greater pain catastrophizing.
Depression | Baseline, 2 weeks post-treatment, 6 week post-treatment
  Change in depression from baseline through 6-week follow-up will be assessed with the Patient Health Questionnaire-2. Scores range from 0 to 6, with higher scores reflecting greater depression.
Anxiety | Baseline, 2 weeks post-treatment, 6 week post-treatment
  Change in anxiety from baseline through 6-week follow-up will be assessed with the Generalized Anxiety Disorder 2-item. Scores range from 0 to 6, with higher scores reflecting greater anxiety.
Prescription Pain Medication Use | Baseline, 2 weeks post-treatment, 6 week post-treatment
  Change in prescription pain medication misuse from baseline through 6-week follow-up will be assessed with the PROMIS Prescription Pain Medication Misuse Short Form. Scores range from 7 to 35, with higher scores reflecting greater medication misuse.
Mindful Pain Management | Baseline, 2 weeks post-treatment, 6 week post-treatment
  Change in the use of mindfulness for pain management from baseline through 6-week follow-up will be assessed with the Mindful Reappraisal of Pain Scale. Scores range from 0 to 54, with higher scores reflecting greater mindful pain management.
Self-Transcendent Experiences | Baseline, 2 weeks post-treatment, 6 week post-treatment
  Change in the the frequency of self-transcendent experiences from baseline through 6-week follow-up will be assessed with the Nondual Awareness Dimensional Assessment. Scores range from 0 to 5, with higher scores reflecting more frequent self-transcendent experiences.

CONTACTS AND LOCATIONS:
Locations (1):
- Brian Science and Symptom Management Center, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No